CLINICAL TRIAL: NCT01130493
Title: A Study to Compare IPX066 and Carbidopa/Levodopa/Entacapone (CLE) Followed by an Open-Label Safety Study of IPX066 in Advanced Parkinson's Disease
Brief Title: A Study to Compare IPX066 and Carbidopa/Levodopa/Entacapone (CLE) Followed by an Open-Label Safety Study of IPX066
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPX066-B09-06
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2017-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination; Stalevo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPX066-CLE-OLE (Other): Dose conversion from CLE to IPX066, IPX066 (Part 1 Period 1), Open-label IPX066, CLE (Part 1 Period 2), OLE (Part 2)
  Interventions: Drug: IPX066; Drug: CLE
- CLE-IPX066-OLE (Other): Dose conversion from CLE to IPX066, CLE (Part 1 Period 1), Open-label IPX066, IPX066 (Part 1 Period 2), OLE (Part 2)
  Interventions: Drug: IPX066; Drug: CLE

INTERVENTIONS:
Drug: IPX066 — experimental product
  Other Names: extended-release carbidopa-levodopa
Drug: CLE — active comparator
  Other Names: carbidopa/levodopa/entacapone

SUMMARY:
This is a study to compare the efficacy of IPX066 and CLE in subjects with advanced Parkinson's disease.

DETAILED DESCRIPTION:
This is a randomized, double-blind, double-dummy, 2 treatment, 2-period crossover study followed by an open-label extension study period.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with idiopathic Parkinson's Disease (PD).
2. At least 30 years old at the time of PD diagnosis.
3. Currently being treated with carbidopa/levodopa/entacapone (CLE) and on a stable regimen of conventional LD for at least 4 weeks and:

   * Requiring a total daily levodopa (LD) dose of at least 400 mg
   * Having a minimum dosing frequency of four times per day.
   * Individual CD-LD or CLE doses that contain an LD dose which is a multiple of 50 mg.
4. Able to differentiate "on" state from "off" state.
5. Have predictable "off" periods.
6. Amantadine, anticholinergics, selective monoamine oxidase (MAO) type B inhibitors (e.g., selegiline, rasagiline) or dopamine agonists are allowed as long as the doses and regimens have been stable for at least 4 weeks prior to Screening and the therapy is intended to be constant throughout the course of the study.
7. Agrees to use a medically acceptable method of contraception throughout the study and for 1 month afterward.

Exclusion Criteria:

1. Diagnosed with atypical Parkinsonism or any known secondary Parkinsonian syndrome.
2. Nonresponsive to LD therapy.
3. Prior functional neurosurgical treatment for PD (e.g., ablation or deep brain stimulation) or if such procedures are anticipated during study participation.
4. Received within 4 weeks of Screening or planning to take during participation in the clinical study: any controlled-release LD product, tolcapone, apomorphine, nonselective MAO inhibitors, or antipsychotics including neuroleptic agents for the purpose of treating psychosis or bipolar disorder.
5. Allergy or hypersensitivity to CD, LD, entacapone, riboflavin, Yellow Dye #5 (tartrazine), citrus fruit or grape juice.
6. History of or currently active psychosis.
7. Active or prior medical conditions such as peptic ulcers or prior surgical (e.g., bowel) procedures that would interfere with LD absorption.
8. Active or history of narrow-angle glaucoma.
9. History of malignant melanoma or a suspicious undiagnosed skin lesion.
10. History of myocardial infarction with residual atrial, nodal, or ventricular arrhythmias, upper gastrointestinal hemorrhage, or neuroleptic malignant syndrome or nontraumatic rhabdomyolysis.
11. Received any investigational medications during the 4 weeks prior to Screening.
12. Unable to swallow large pills (e.g., large vitamin pills).
13. Pregnant or breastfeeding.
14. Subjects who are unable to complete a symptom diary.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Impax Study Director, Study Director — Impax Laboratories, LLC
Locations (24):
- United States (12):
  - Margolin Brain Institute, Fresno, California
  - The Parkinson's Institute in Sunnyvale, Sunnyvale, California
  - UM Movement Disorders Center, Miami, Florida
  - Charlotte Neurological Services, Port Charlotte, Florida
  - USF Parkinson's and Movement Disorders Center, Tampa, Florida
  - Quest Research Institute, Bingham Farms, Michigan
  - University Health Systems, Las Vegas, Nevada
  - Parkinson's Disease and Movement Disorders Center of Long Island, Commack, New York
  - Kingston Neurological Associates, Kingston, New York
  - University Neurology, Inc, Cincinnati, Ohio
  - Sentara Neurological Associates, Virginia Beach, Virginia
  - Booth Gardner Parkinson's Care Center, Kirkland, Washington
- France (2):
  - Hôpital Gabriel Montpied-Service de Neurologie A-, Clermont-Ferrand
  - Service de neurologie-Hôpital de la Timone-, Marseille
- Germany (5):
  - Praxis für Neurologie, Psychiatrie und Psychotherapie Achim, Achim
  - Praxis Dres. Bitter/Schumann, Bochum
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Klinik für Neurologie, Stadtroda, Stadtroda
  - RKU, Neurologische Klinik der Universität Ulm, Ulm
- Italy (5):
  - Casa di Cura Villa Margherita, Arcugnano
  - San Raffaele Cassino, San Raffaele Cassino,, Cassino
  - Dipartimento di Oncologia e Neuroscienze, Università G. D'Annunzio, Chieti
  - Ospedale della Misericordia, Grosseto
  - IRCCS San Raffaele Pisana, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morgan JC, Dhall R, Rubens R, Khanna S, Gupta S. Dosing Patterns during Conversion to IPX066, Extended-Release Carbidopa-Levodopa (ER CD-LD), in Parkinson's Disease with Motor Fluctuations. Parkinsons Dis. 2018 Oct 22;2018:9763057. doi: 10.1155/2018/9763057. eCollection 2018. PMID 30425824

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date first patient enrolled: March 22, 2011 Date last patient completed: January 12, 2012
Pre-assignment Details: Following enrollment, all subjects were converted from stable doses of CLE to IPX066 prior to randomization. Following dose conversion, subjects were randomized into one of the two treatment sequences.
Groups:
- IPX066 Conversion: All subjects were converted to IPX066 during an open-label period
- IPX066-Open-label IPX066 Washout-CLE-OLE: IPX066 (Per Protocol: Part 1 Period 1), Open-label washout IPX066, CLE (Per Protocol: Part 1 Period 2), OLE (Per Protocol: Part 2)
- CLE-Open Label IPX066 Washout-IPX066-OLE: CLE (Per Protocol: Part 1 Period 1), Open-label washout IPX066, IPX066 (Per Protocol: Part 1 Period 2), OLE (Per Protocol: Part 2)
Period: Open-label Dose Conversion to IPX066
Arm/Group | IPX066 Conversion | IPX066-Open-label IPX066 Washout-CLE-OLE | CLE-Open Label IPX066 Washout-IPX066-OLE
Started | 110 (During the open-label dose conversion to IPX066, all subjects received IPX066) | 0 | 0
Completed | 91 | 0 | 0
Not Completed | 19 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 0
Not completed — Lack of Efficacy | 7 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 0
Not completed — Diary imcomplete | 1 | 0 | 0
Period: Part 1: Double-blind Treatment Period 1
Arm/Group | IPX066 Conversion | IPX066-Open-label IPX066 Washout-CLE-OLE | CLE-Open Label IPX066 Washout-IPX066-OLE
Started | 0 (91 subjects completed IPX066 dose conversion and were then randomized to the two treatment sequences) | 48 (48 were randomized to IPX066-CLE double-blind treatment sequence) | 43 (43 were randomized to CLE-IPX066 double-blind treatment sequence)
Completed | 0 | 46 | 43
Not Completed | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0
Period: Part 1: Open-Label IPX066 Washout
Arm/Group | IPX066 Conversion | IPX066-Open-label IPX066 Washout-CLE-OLE | CLE-Open Label IPX066 Washout-IPX066-OLE
Started | 0 | 46 | 43
Completed | 0 | 45 | 41
Not Completed | 0 | 1 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Part 1: Double-blind Treatment Period 2
Arm/Group | IPX066 Conversion | IPX066-Open-label IPX066 Washout-CLE-OLE | CLE-Open Label IPX066 Washout-IPX066-OLE
Started | 0 | 45 | 41
Completed | 0 | 45 | 39
Not Completed | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Noncompliance | 0 | 0 | 1
Period: Part 2: OLE
Arm/Group | IPX066 Conversion | IPX066-Open-label IPX066 Washout-CLE-OLE | CLE-Open Label IPX066 Washout-IPX066-OLE
Started (10 subjects did not roll over to Part 2 (OLE) as it was optional. Reasons were not collected.) | 0 | 39 (All subjects received IPX066 during OLE) | 35 (No subjects received CLE during OLE)
Completed | 0 | 36 | 30
Not Completed | 0 | 3 | 5
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Participants who completed the Dose Conversion period and were randomized into the double-blind crossover portion of the study.
Groups:
- All Study Participants: Participants who were randomized to receive either IPX066 or IR CD-LD in Part 1 of the study and then IPX066 in Part 2 (open-label extension).
Arm/Group | All Study Participants
Number analyzed (Participants) | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 79
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 89
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 44
  Italy | 26
  Germany | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of "OFF" Time During Waking Hours
Description: Using a Parkinson's disease diary, subjects recorded a state of "asleep", "OFF", "ON without dyskinesia," "ON with non-troublesome dyskinesia," or "ON with troublesome dyskinesia" every 30 minutes over a 24-hour day for the last 3 days of each double-blind crossover treatment period.
  Mean percentage of "OFF" Time During Waking Hours was calculated. "Off" Time is Time when medication has worn off and is no longer providing benefit with regard to mobility, slowness, and stiffness.
Time Frame: 3 days of data immediately prior to the end of each 2 week treatment period
Population: Participants who completed both treatment periods and completed PD diary for both Period 1 and Period 2
Measure: Mean (Standard Deviation); unit: Percent
Groups:
- IPX066: Participants who received IPX066 in either Period 1 or Period 2
- CLE (Active Comparator): Participants who received CLE in either Period 1 or Period 2
Arm/Group | IPX066 | CLE (Active Comparator)
Number analyzed (Participants) | 83 | 83
Percent | 23.98 (16.242) | 32.48 (21.917)

2. Secondary Outcome: Total "OFF" Time During Waking Hours
Description: Using a Parkinson's disease diary, subjects recorded a state of "asleep", "OFF", "ON without dyskinesia," "ON with non-troublesome dyskinesia," or "ON with troublesome dyskinesia" every 30 minutes over a 24-hour day for the last 3 days of each double-blind crossover treatment period.
  Mean Total "Off" Time During Waking Hours was calculated. "Off" Time is Time when medication has worn off and is no longer providing benefit with regard to mobility, slowness, and stiffness.
Time Frame: 3 days of data immediately prior to the end of each 2 week treatment period
Population: Participants who completed both treatment periods and completed PD diary for both Period 1 and Period 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IPX066 | CLE (Active Comparator)
Number analyzed (Participants) | 83 | 83
hours | 3.82 (2.558) | 5.22 (3.672)

3. Secondary Outcome: Total "On" With No Troublesome Dyskinesia
Description: Using a Parkinson's disease diary, subjects recorded a state of "asleep", "OFF", "ON without dyskinesia," "ON with non-troublesome dyskinesia," or "ON with troublesome dyskinesia" every 30 minutes over a 24-hour day for the last 3 days of each double-blind crossover treatment period.
  Mean Total "On" with No Troublesome Dyskinesia was calculated. "On" Time is when medication is providing benefit with regard to mobility, slowness, and stiffness.
Time Frame: 3 days of data immediately prior to the end of each 2 week treatment period
Population: Participants who completed both treatment periods and completed PD diary for both Period 1 and Period 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IPX066 | CLE (Active Comparator)
Number analyzed (Participants) | 83 | 83
hours | 11.36 (3.259) | 9.98 (3.764)

4. Secondary Outcome: UPDRS Part II Plus Part III
Description: Unified Parkinson's Disease Rating Scale (UPDRS) Part II (Activities of Daily Living) and Part III (Motor Examination). Part II consists of 14 questions, each ranges from 0 (Normal/None) - 4 (Worst) with a total score of 0 - 72. Part III consists of 27 questions, each ranges from 0 (Normal/None) - 4 (Worst) with a total score of 0 - 108.
  The UPDRS Part II Plus Part III scores ranged from 0 (no problems with daily living or mobility) to 180 (severe problems with daily living and mobility.
Time Frame: End of each double-blind treatment period.
Population: Participants who completed both treatment periods
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | IPX066 | CLE (Active Comparator)
Number analyzed (Participants) | 84 | 84
Scores on a scale | 29.3 (15.02) | 31.7 (14.89)

5. Secondary Outcome: Subject Preference
Description: Subjects who completed both treatments were asked to indicate a preference for Treatment Period 1 or Treatment Period 2 or no preference. Preferences for a particular treatment period were mapped to the associated treatment and reported.
Time Frame: End of Study (week 11)
Population: Participants who completed both treatment periods
Measure: Count of Participants; unit: Participants
Groups:
- Number of Participants Who Preferred IPX066: Participants who completed both treatment periods and who had a preference for IPX066
- Number of Participants Who Preferred CLE: Participants who completed both treatment periods and who had a preference for CLE
- Number of Participants Who Had no Preference: Participants who completed both treatment periods and who did not indicate a preference for either treatment
Arm/Group | Number of Participants Who Preferred IPX066 | Number of Participants Who Preferred CLE | Number of Participants Who Had no Preference
Number analyzed (Participants) | 84 | 84 | 84
Participants | 44 | 23 | 17

ADVERSE EVENTS:
Groups:
- Dose Conversion: Participants were to be converted from stable doses of CLE to open-label IPX066 over a 6-week period
- IPX066: Participants first received 2 weeks of IPX066 followed by an approximate 7-day washout period of IPX066 treatment followed by another 2 weeks of CLE.
- CLE (Active Comparator): Participants first received 2 weeks of CLE followed by an approximate 7-day washout period of IPX066 treatment followed by another 2 weeks of IPX066.
- Washout: Participants receive open-label IPX066 for 1 week
Arm/Group | Dose Conversion | IPX066 | CLE (Active Comparator) | Washout
Serious Adverse Events (participants affected / at risk) | 2/91 | 1/89 | 0/88 | 1/89
Other Adverse Events (participants affected / at risk) | 14/91 | 13/89 | 2/88 | 1/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Conversion (N=91) | IPX066 (N=89) | CLE (Active Comparator) (N=88) | Washout (N=89)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Toxicity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Conversion (N=91) | IPX066 (N=89) | CLE (Active Comparator) (N=88) | Washout (N=89)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No